CLINICAL TRIAL: NCT03455335
Title: A Phase 1b, Open Label, Uncontrolled, Non-randomized Dose-escalation Study to Examine the Safety of Intramuscular Autologous Transplantation of Escalating Doses of Mesenchymal Stem Cells to Patients With no Option Critical Limb Ischemia.
Brief Title: Autologous Stem Cells for the Treatment of No Option Critical Limb Ischemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Professor Tim O Brien, Professor Tim o Brien, National University of Ireland, Galway, Ireland
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013-001
Record Dates: First submitted 2018-02-16; First posted 2018-03-06 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Advanced Therapeutic Medicinal Product ( ATMP) Bone Marrow Derived Mesenchymal Stem Cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose cohort (Experimental): 20 million hMSCs .
  Interventions: Drug: 20 million hMSCs
- mid dose cohort (Experimental): 40 million hMSCs
  Interventions: Drug: 40 million hMSCs
- high dose cohort (Experimental): 80 million hMSCs .
  Interventions: Drug: 80 million hMSCs

INTERVENTIONS:
Drug: 20 million hMSCs
  Other Names: 20 million hMSCs intramuscularly
  Arms: low dose cohort
Drug: 40 million hMSCs
  Other Names: 40 million hMSCs intramuscularly
  Arms: mid dose cohort
Drug: 80 million hMSCs
  Other Names: 80 million hMSCs intramuscularly
  Arms: high dose cohort

SUMMARY:
The trial is a phase 1b, open label, uncontrolled, non-randomized dose-escalation study of autologous bone marrow-derived MSCs. Following informed consent, patients who meet the criteria will be screened and enrolled. Up to 100 mls of bone marrow will be harvested from the participant from which MSCs will be culture expanded. In this dose escalation study, 3 participants on each cohort will be treated with a targeted dose of either 20 million hMSC; 40 million hMSC; or 80 million hMSC. The cells will be administered to the ischemic leg by 20 intramuscular injections of approximately 0.5ml per injection . Treatment groups will be completed sequentially, beginning with the lowest dose group.

DETAILED DESCRIPTION:
This is a phase 1b, open label, uncontrolled, non-randomized dose-escalation study to examine the safety of intramuscular autologous transplantation of escalating doses of mesenchymal stem cells to patients with no option critical limb ischemia.

Trial Aims and Objectives: To examine the safety of intramuscular transplantation of escalating doses of autologous bone marrow derived mesenchymal stem cells to patients with no option critical limb ischemia.

Patient Population: Patients with critical limb ischemia who are not candidates for revascularization.

Trial Setting:HRB Clinical Research Facility Galway and Galway University Hospitals.

Trial Intervention:Intramuscular delivery of autologous bone marrow-derived mesenchymal stem cells to patients with no option critical limb ischemia.

Study Design: Open label, uncontrolled, non-randomized, dose escalation study. Sample Size: 9 Method of Participant Assignment:Sequential administration of 3 escalating doses of autologous bone marrow-derived mesenchymal stem cells.

Examination Points: Day 0, 7, 30, 90, 180, 365 and 730 Primary Outcome: Serious adverse events that are attributable to intervention. Secondary Outcomes :Amputation free survival, median time to amputation, TcPo2, ABI, pain scale, ulcer healing, quality of life assessments, collateral vessel formation detected by MRI at 12 months.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled into the study

1. Men and women between the ages of 18 and 85
2. Voluntary written informed consent, given before performance of any study-related procedure not part of standard medical care, and with the understanding that consent may be withdrawn at any time without prejudice to future medical care
3. Presented with CLI with rest pain or ulceration with no option for revascularization agreed by an expert panel including an interventional radiologist and vascular surgeon; CLI defined as persistent ischemic rest pain for greater than or equal to 2 weeks and/or ulceration or gangrene of the toe or foot
4. Estimated life expectancy > 6 months as deemed by patient's clinician and/or investigator
5. Suitable candidate for a bone marrow aspiration, deemed by Consultant Haematologist
6. Chronic critical limb ischaemia with rest pain (Rutherford Class 4) or mild-to-moderate tissue loss (Rutherford Class 5) who are not candidates for revascularisation
7. Medically fit to undergo bone marrow harvest and stem cell intramuscular injection
8. One of the following haemodynamic parameters: ankle systolic pressure < 70 mmHg or ABI <0.9 TBI <0 .6 TcPO2 <60mmHg on room air

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Has received prior therapy with MSCs
2. Has had previous amputation of the talus or above
3. Has failed revascularization within 2 weeks before entry to the study
4. Known Aortoiliac disease with > 50% stenosis
5. Contraindication to intramuscular procedure, including active infection in the affected limb, or wet gangrene or exposed bone or tendon in lower limb with CLI, or in the opinion of the attending clinician, is unsuitable for intramuscular procedure
6. Severe co-morbidity limiting 6 month survival of patients
7. Abnormal liver function as defined by AST and ALT > 2.5 fold the ULN and total bilirubin > 1.5 ULN
8. Significant cognitive impairment (Mini Mental Status Examination <22)
9. Presence of proliferative retinopathy (in participants with diabetes mellitus only)
10. Presence of poorly controlled diabetes mellitus with HbAIc > 10% within previous 3 months
11. HIV or HBsAg positive
12. Presence of acute coronary syndrome
13. Patient has known active malignancy
14. Pregnancy
15. Likely inability to comply with the protocol or cooperate fully with the investigator and site personnel
16. Patient taking other investigational drugs at the time of enrolment or within 28 days of enrolment
17. Rutherford class 6 CLI
18. Significant bone marrow dysfunction, based on assessment by Haematologist or an established diagnosis of myelodysplasia, or myeloproliferative disorder etc.
19. Bleeding diathesis, coagulopathy, thrombocytopenia etc.
20. Patients in whom delay incurred by attempts at limb salvage using MSCs will adversely affect prognosis in the opinion of the responsible attending clinician
21. Patients with known allergy to foetal bovine serum or trypsin

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
The number of Serious Adverse Events that are attributable to the treatment | 12 months
  The number of Serious Adverse Events that are attributable to the MScs
The severity of Serious Adverse Events that are attributable to the treatment | 12 months
  The number of Serious Adverse Events that are attributable to the MScs

SECONDARY OUTCOMES:
Amputation free survival | 12 months
  Efficacy measured by the presence or absence of the target limb
median time to amputation, | 12 months
  Efficacy measured by the duration from time of cell administration to time of amputation if applicable.
Change in Transcutaneous Pressure of Oxygen TcPO2 | 12 months
  Efficacy will be determined by improvement from baseline in mmHg
Change in Ankle Brachial Index | 12 months
  "Ankle Brachial Index: An indicator of peripheral perfusion measured by dividing Ankle Pressure (mmHg) by brachial pressure (mmHg) (normal ABI is 1.0 ). Efficacy outcome will be measured by improvement from baseline . The higher the ABI, the better the outcome."
Collateral vessel formation | 12 months
  Efficacy will be determined the presence of collateral vessel formation as detected by MRI
Change in Ischemic rest pain | 12 months.
  Efficacy will be determined by decrease in score from baseline as measured by verbal analogue scale (0 = no pain, 10 = worst pain in life)
Change in Ulcer size | 12 months.
  Efficacy will be determined by decrease in the surface area from baseline as measured by ImageJ software and or complete healing of the ulcer
Change in Quality of Life | 12 months.
  Efficacy will be measured using the EQ 5D Quality of Life assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: Timothy O Brien, PhD, Principal Investigator — NUIG
Locations (1):
- Galway University Hospital, Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohamed SA, Howard L, McInerney V, Hayat A, Krawczyk J, Naughton S, Finnerty A, Holohan M, Duffy A, Moloney T, Kavanagh E, Burke P, Liew A, Tubassam M, Walsh SR, O'Brien T. Autologous bone marrow mesenchymal stromal cell therapy for "no-option" critical limb ischemia is limited by karyotype abnormalities. Cytotherapy. 2020 Jun;22(6):313-321. doi: 10.1016/j.jcyt.2020.02.007. Epub 2020 Apr 6. PMID 32273232
- [Background] EU Clinical Trials Register Clinical trial results 2013-003447-37 version 1 EU-CTR publication date: of 21 01 January 2021